CLINICAL TRIAL: NCT00926692
Title: Investigations Regarding B-cell Subsets in Humans
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Daniel Griffin, Fellow Infectious Diseases, Northwell Health
Other Study IDs: GCRC 0266
Record Dates: First submitted 2009-06-19; First posted 2009-06-23 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: B-cells; CD5+; B1 Cells; Healthy Controls
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy Subjects: All subjects are considered healthy
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — Subject will have blood draw.

SUMMARY:
The aim of this research is to define the human equivalent of mouse B1 cells.

DETAILED DESCRIPTION:
The specific aim of this research project is to define the human equivalent of mouse B1 cells. This will be done by evaluating IgM secretion, surface markers, functional characteristics, V gene usage, N-region addition, and phosphorylation status of intracellular proteins, gene expression, sequencing of immunoglobulin genes, determination of antigenic specificity, replication history, and response to different stimuli.

The goal of this project is to begin to the translation of decades of basic science research and research in the mouse model into the human system. It is believed that properly defining this B cell subset in humans will lead to better therapeutics, prognostics and prevention for a number of disease including infections, autoimmune disease, and cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subject is considered by the physician to be a healthy adult.

Exclusion Criteria:

* Subject is under the age of 18
* Subject has an infection or is currently ill

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Control Population
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2009-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Presence of B-1 cells in humans | determined over the years study in effect
  an equivalent cell type was isolated in humans

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Griffin, M.D., Principal Investigator — Feinstein Institute for Medical Research
Locations (1):
- Feinstein Institute for Medical Research, Manhasset, New York, United States